CLINICAL TRIAL: NCT04213950
Title: Improving Adherence to Rabies Postexposure Prophylaxis Guideline Recommendations for Rabies Immune Globulin at a Multi-hospital Health System Through Education, Collaboration, and Clinical Decision Support
Brief Title: Improving Adherence to Rabies PEP Guideline Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Joshua Swan, PharmD, MPH, FCCM, Associate Professor of Pharmacy in Surgery and Outcomes Research, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00022539
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Rabies; Rabies Human; Rabies Virus Infection
Keywords: rabies immune globulin; rabies vaccine; rabies postexposure prophylaxis; rabies PEP; rabies IG
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Intervention Model Description: The study consists of 2 groups: (1) the historical control group and (2) the post-implementation group. The historical control group includes patients who received rabies PEP from January 2015 to June 2018. The quality improvement bundle will be implemented across the Houston Methodist health system in December 2019. The post-implementation group includes patients who receive rabies PEP within 12 months following bundle implementation. An estimated sample size of 70 patients in the post-implementation group and 254 patients in the historical control group will provide 80% power to detect an absolute increase of 20% in the primary endpoint using a two-sided alpha of 0.05.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-implementation group (Experimental): The post-implementation group will receive care that is enhanced by the rabies PEP quality improvement bundle.
  Interventions: Other: Rabies PEP quality improvement bundle
- Historical control group (No Intervention): The historical control group received care prior to implementation of the quality improvement bundle.

INTERVENTIONS:
Other: Rabies PEP quality improvement bundle — The rabies PEP quality improvement bundle consists of (1) electronic health record enhancements to support rabies PEP treatment selection, administration, and discharge process; (2) education to ED staff on rabies PEP; and (3) education to patients on rabies PEP and follow-up care.
  Arms: Post-implementation group

SUMMARY:
This quasi-experimental, quality improvement study will be conducted across the Houston Methodist system, including all hospital-based and freestanding emergency departments (ED). Previous research identified opportunities to improve patient selection and delivery of rabies immune globulin (IG) as recommended by Centers for Disease Control and Prevention (CDC) guideline recommendations for rabies postexposure prophylaxis (PEP). The purpose of this study is to develop, implement, and measure the impact of a quality improvement bundle that consists of (1) rabies PEP electronic health records (EHR) enhancements, (2) education to ED staff, and (3) education to patients. Adherence to quality indicators, which are based on CDC guideline recommendations, for patient selection and delivery of rabies IG for 12 months following implementation (post-implementation group) will be compared with a historical control group.

DETAILED DESCRIPTION:
BACKGROUND: Rabies infection can occur in humans when key elements of the rabies PEP regimens are omitted or incorrectly administered. The CDC Advisory Committee on Immunization Practices (ACIP) recommends that patients who are exposed to rabies virus should receive prompt and thorough wound cleansing followed by administration of human rabies IG and rabies vaccine. Previous research identified three opportunities to improve adherence to CDC guideline recommendations for rabies PEP: (1) infiltration of rabies IG into and around the wounds, if anatomically feasible, (2) administration of rabies IG at an anatomical site distant from rabies vaccine administration, and (3) avoiding administration of rabies IG into the buttock.

STUDY DESIGN: This quasi-experimental, quality improvement study evaluates adherence to 6 quality indicators, which are based on CDC guideline recommendations, for patient selection and delivery of rabies IG before and after implementation of the rabies PEP quality improvement bundle. The quality improvement bundle includes EHR enhancements, ED staff education, and patient education. Patients who receive at least one dose of rabies IG or rabies vaccine at a study site during the study period will be included in this study. The historical control group includes patients treated prior to bundle implementation. The post-implementation group includes patients treated within 12 months following bundle implementation. The primary outcome is full adherence to all 6 quality indicators for rabies IG selection and delivery.

ELIGIBILITY:
Inclusion Criteria:

• Receive at least one dose of rabies IG or rabies vaccine at a study site during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-29 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Full adherence to 6 quality indicators for rabies immune globulin patient selection and delivery | 1 day; during the patient's first medical encounter at a study site for rabies PEP
  The proportion of patients who achieve full adherence to a composite of all 6 quality indicators for rabies IG patient selection and delivery: (1) appropriate patient selection, (2) appropriate dose, (3) appropriate timing, (4) administration into and around the wound if anatomically feasible, (5) administration distant from rabies vaccine, and (6) administration that avoids the buttock (unless the wound is near the buttock) among patients who received rabies PEP.

SECONDARY OUTCOMES:
Adherence to each of the 6 quality indicators for rabies immune globulin patient selection and delivery | 1 day; during the patient's first medical encounter at a study site for rabies PEP
  The proportion of patients who achieve adherence to each of the 6 quality indicators for rabies IG patient selection and delivery.
Volume of rabies immune globulin administered into or around wounds | 1 day; during the patient's first medical encounter at a study site where rabies IG is administered
  The mean percent of the total volume of rabies IG administered into or around wounds, if anatomically feasible.
Clear documentation of rabies immune globulin administration site | 1 day; during the patient's first medical encounter at a study site where rabies IG is administered
  The proportion of patients with clear EHR documentation of rabies IG administration sites
Incidence of compartment syndrome | For 7 days following rabies IG administration
  The incidence of compartment syndrome at a rabies IG infiltration site that was documented in the EHR within 7 days of rabies IG administration
Incidence of sciatic nerve injury | For 21 days following rabies IG administration
  The incidence of sciatic nerve injury that was documented in the EHR within 21 days of rabies IG administration among patients who receive rabies IG into the buttock

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Swan, PharmD, MPH, Principal Investigator — Houston Methodist Health System
Locations (15):
- United States (15):
  - Houston Methodist Emergency Department at Baytown, Baytown, Texas
  - Houston Methodist Emergency Care Center in Cypress, Cypress, Texas
  - Houston Methodist Hospital Emergency Department, Houston, Texas
  - Houston Methodist Emergency Care Center at Voss, Houston, Texas
  - Houston Methodist Emergency Department at Willowbrook Hospital, Houston, Texas
  - Houston Methodist Emergency Department at West, Houston, Texas
  - Houston Methodist Emergency Care Center at Kirby, Houston, Texas
  - Houston Methodist Emergency Care Center in Sienna Plantation, Missouri City, Texas
  - Houston Methodist Emergency Department at Clear Lake, Nassau Bay, Texas
  - Houston Methodist Emergency Care Center in Pearland, Pearland, Texas
  - Houston Methodist Emergency Care Center in Cinco Ranch, Richmond, Texas
  - Houston Methodist Emergency Care Center in Spring, Spring, Texas
  - Houston Methodist Emergency Department at Sugar Land, Sugar Land, Texas
  - Houston Methodist Emergency Care Center in The Woodlands, The Woodlands, Texas
  - Houston Methodist Emergency Department at The Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang GS, Rizk E, Bui LN, Iso T, Sartain EI, Tran AT, Swan JT. Adherence to guideline recommendations for human rabies immune globulin patient selection, dosing, timing, and anatomical site of administration in rabies postexposure prophylaxis. Hum Vaccin Immunother. 2020;16(1):51-60. doi: 10.1080/21645515.2019.1632680. Epub 2019 Aug 1. PMID 31210569
- [Background] Rupprecht CE, Briggs D, Brown CM, Franka R, Katz SL, Kerr HD, Lett SM, Levis R, Meltzer MI, Schaffner W, Cieslak PR; Centers for Disease Control and Prevention (CDC). Use of a reduced (4-dose) vaccine schedule for postexposure prophylaxis to prevent human rabies: recommendations of the advisory committee on immunization practices. MMWR Recomm Rep. 2010 Mar 19;59(RR-2):1-9. PMID 20300058
- [Background] Bharti OK, Madhusudana SN, Gaunta PL, Belludi AY. Local infiltration of rabies immunoglobulins without systemic intramuscular administration: An alternative cost effective approach for passive immunization against rabies. Hum Vaccin Immunother. 2016 Mar 3;12(3):837-42. doi: 10.1080/21645515.2015.1085142. PMID 26317441
- [Background] Bharti OK, Madhusudana SN, Wilde H. Injecting rabies immunoglobulin (RIG) into wounds only: A significant saving of lives and costly RIG. Hum Vaccin Immunother. 2017 Apr 3;13(4):762-765. doi: 10.1080/21645515.2016.1255834. Epub 2017 Feb 22. PMID 28277089
- [Background] Wilde H, Sirikawin S, Sabcharoen A, Kingnate D, Tantawichien T, Harischandra PA, Chaiyabutr N, de Silva DG, Fernando L, Liyanage JB, Sitprija V. Failure of postexposure treatment of rabies in children. Clin Infect Dis. 1996 Feb;22(2):228-32. doi: 10.1093/clinids/22.2.228. PMID 8838177
- [Background] Madhusudana SN, Aggarwal P, Tripathi KK. Failure of rabies postexposure treatment with purified chick embryo cell (PCEC) vaccine. Vaccine. 1989 Oct;7(5):478-9. doi: 10.1016/0264-410x(89)90185-0. No abstract available. PMID 2815983
- [Background] Jung Kim H, Hyun Park S. Sciatic nerve injection injury. J Int Med Res. 2014 Aug;42(4):887-97. doi: 10.1177/0300060514531924. Epub 2014 Jun 11. PMID 24920643
- [Background] National Center for Immunization and Respiratory Diseases. General recommendations on immunization --- recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2011 Jan 28;60(2):1-64. PMID 21293327
- [Background] HyperRab® [rabies immune globulin (human)] [package insert]. Grifols Therapeutics Inc., Research Triangle Park, NC, USA. 2018.
- [Background] Salva EP, Dimaano EM, Villarama JB, Suquilla JT. An evaluation of the safety and potency of equine rabies immunoglobulin through measurements of suppression on vaccine induced antibody production among healthy volunteers. Philippine Journal of Internal Medicine. 2014;52(2):1-7.
- [Background] HyperRab® S/D (rabies immune globulin [human]) [package insert]. Grifols Therapeutics Inc., Clayton, NC. 2012.
- [Background] Kline DG, Kim D, Midha R, Harsh C, Tiel R. Management and results of sciatic nerve injuries: a 24-year experience. J Neurosurg. 1998 Jul;89(1):13-23. doi: 10.3171/jns.1998.89.1.0013. PMID 9647167
- [Background] GILLES FH, FRENCH JH. Postinjection sciatic nerve palsies in infants and children. J Pediatr. 1961 Feb;58:195-204. doi: 10.1016/s0022-3476(61)80158-3. No abstract available. PMID 13705320
- [Background] Bergeson PS, Singer SA, Kaplan AM. Intramuscular injections in children. Pediatrics. 1982 Dec;70(6):944-8. PMID 6755373
- [Background] Centers for Disease Control and Prevention. Human Rabies. 2017; https://www.cdc.gov/rabies/location/usa/surveillance/human_rabies.html. Accessed Jan 10, 2019.